CLINICAL TRIAL: NCT03711565
Title: Oscillatory Versus Non-Oscillatory Nasal Continuous Airway Pressure Neonatal Respiratory Support
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The research equipment was not available for more than a year after the study was submitted. A new trial was being done during delivery of patients that competed with the study.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 828375
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Neonatal Respiratory Distress Related Conditions
Keywords: Nasal CPAP; High Frequency NCPAP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Regular Nasal CPAP using a conventional ventilator (Active Comparator): Regular nasal CPAP for management of respiratory distress Patient will have regular nasal CPAP placed via nasal prongs with level of pressure adjusted and level of oxygen adjusted as needed for acceptable oxygenation and ventilation
  Interventions: Device: Regular Nasal CPAP using a conventional ventilator
- High Frequency Nasal CPAP (Active Comparator): High Frequency Nasal CPAP for management of respiratory distress Patient will be connected to the high frequency device through nasal prongs. The pressure, frequency and amplitude of the pulsations will be adjusted as needed to provide acceptable oxygenation and ventilation
  Interventions: Device: High Frequency Nasal CPAP

INTERVENTIONS:
Device: Regular Nasal CPAP using a conventional ventilator — The Nasal CPAP is connected to the patient via prongs in the nose. Pressure adjustments are made to improve lung inflation. The frequency and pressure can be adjusted as needed to improve the patient's oxygen and carbon dioxide levels
  Arms: Regular Nasal CPAP using a conventional ventilator
Device: High Frequency Nasal CPAP — High Frequency Nasal CPAP for management of respiratory distress Patient will be connected to the high frequency device through nasal prongs. The Bronchotron produces a pressure that is variable with an adjustable frequency that is equal or greater than 500 times per minute connecting to prongs in the patient's nose. The pressure, frequency and amplitude of the pulsations will be adjusted as needed to provide acceptable oxygenation and ventilation.
  Arms: High Frequency Nasal CPAP

SUMMARY:
Controlled randomized trial looking at Standard nasal continuous airway pressure (CPAP) respiratory support versus High Frequency CPAP in neonates who require respiratory support or who are being extubated and require support post extubation. Patients will be evaluated for need to be reintubated and oxygen requirement and PaCO2 levels

DETAILED DESCRIPTION:
This study is a randomized controlled trial comparing High Frequency nasal CPAP versus standard nasal CPAP. The patient population includes preterm newborns who require respiratory support but do not need to be initially intubated and preterm or term infants who are being extubated and will require support for the continued lung disease. After obtaining parental consent the patient will be randomized to one of the two treatments. Patients will be followed for requirement of level of oxygen and blood gases looking at acidity (pH) and PaCO2 and Bicarbonate(HCO3). A respiratory index score will be measured. Attending physician will determine the need for the patient to be intubated or reintubated depending on the patient selected. Additionally, frequency, duration and severity of Apnea, Bradycardia and Desaturation events will be recorded. Also safety issues to include pulmonary airleak, nasal injury, facial edema and scalp edema due to straps holding the device in place will be recorded. Also gaseous distension of the stomach and intestines will be assessed and compared between treatment arms. This study is not powered to look at long term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Newborn (0-28 days of age) admitted to Neonatal Intensive care unit (NICU)
* Ordered Respiratory treatment of Nasal Continuous Airway Pressure (NCPAP) respiratory support

Exclusion Criteria:

* Major congenital defect
* Known or suspected chromosomal disorder

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Respiratory Index Score (RSI) | 72 hours after initiation of support
  The scale is scored based on Fio2 (0 = <30%, 1 = 30-39%, 2 = 40-49%, 3 = > or equal to 50%), CPAP/Paw (0 = <6, 1 = 6-7, 2 = 7-8, 3 = >8), Spontaneous Respiratory Rate(RR) (0 = <40, 1 = 40-59, 2 = 60-79, 3 = > or equal to 80), Retractions (0 = none, 1 = mild, 2 = moderate, 3 = severe), and Apnea (0 = none, 1 = 1/2/2015, 2 = 3/4/2015, 3 = >4). Average index scores will be compared between conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Health, Sacramento, California, United States